CLINICAL TRIAL: NCT02126735
Title: Metabolic and Cardiovascular Impact of CD36 Deficiency in African Americans
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cyndya Shibao, Assistant Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: 121525
Record Dates: First submitted 2013-10-14; First posted 2014-04-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, white cells
Oversight: Data Monitoring Committee: No

SUMMARY:
CD36, a protein that facilitates tissue uptake of fat, as a common link between blood fat concentrations and metabolic disease states such as diabetes mellitus. Genetic variants in the CD36 gene are more common in African Americans compared to Whites and it may confer protection against metabolic diseases by altering the amount of fat in the blood.

The purpose of this study is to compare the levels of fat in the blood and to assess endothelial dysfunction among carriers versus non-carriers of the coding SNP, rs3211938 of the CD36 gene after a high fat meal challenge

ELIGIBILITY:
Inclusion Criteria:

* African American men and women age 18-65 years of age
* BMI 25-45 kg/m2

Exclusion Criteria:

* Diabetes
* Pregnancy
* Use of nicotinic acid for dyslipidemia
* History of nutrient malabsorption
* Clinically significant hepatic or renal disease, OR serum creatinine or liver function tests > 2times upper limits of normal
* Symptomatic acute or chronic gallbladder disease
* Any underlying or acute disease requiring regular medication which could in the principal investigator's opinion possibly pose a threat to the subject or make implementation of the protocol difficult
* Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
* Patient unwilling or unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: we will recruit subjects locally
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve triglycerides levels after high fat meal | Baseline values prior to high fat meal and at 10, 20, 30, 60, 120, 240 & 360 minutes
  We expect that subjects heterozygous for the minor allele of CD36 rs3211938 (G/T) would have an increase of 250 units in the area under the curve for triglycerides which is ~50% of the observed difference between patients with CD36 deficiency and normal controls. Assuming that the common standard deviation is 199, using a two group t-test with a type I error of 0.05, a total of 28 subjects (14 carriers and 14 non-carriers) would provide 90% power to detect a difference in our primary endpoint between carriers versus non-carriers of genotype

SECONDARY OUTCOMES:
percent change in flow mediated dilation at baseline and 4 hours after a high fat meal | Change from baseline in flow mediated dilation at 4 hours after high fal meal
  our primary outcome will be the percent change in flow mediated dilation at baseline and 4 hours after a high fat meal (peak effect). Assuming a conservative estimate of standard deviation of 3.19 our proposed study with a total of 28 subjects (14 carriers and 14 non-carriers) would have at least 80% power with type I error of 0.05 to detect a minimum difference in the mean response of 3.5 %.

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya A Shibao, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shibao CA, Celedonio JE, Tamboli R, Sidani R, Love-Gregory L, Pietka T, Xiong Y, Wei Y, Abumrad NN, Abumrad NA, Flynn CR. CD36 Modulates Fasting and Preabsorptive Hormone and Bile Acid Levels. J Clin Endocrinol Metab. 2018 May 1;103(5):1856-1866. doi: 10.1210/jc.2017-01982. PMID 29546316
- [Derived] Marinos A, Celedonio JE, Ramirez CE, Gottlieb J, Gamboa A, Hui N, Yu C, Stein CM, Biaggioni I, Shibao CA. Time-Course Analysis of Flow Mediated Dilation for the Evaluation of Endothelial Function After a High-Fat Meal in African Americans. J Am Heart Assoc. 2015 Nov 5;4(11):e002388. doi: 10.1161/JAHA.115.002388. PMID 26541392